CLINICAL TRIAL: NCT03774394
Title: Impact of Chronic Kidney Disease (CKD) on Pharmacodynamic Profiles of the P2Y12 Receptor Inhibitor Clopidogrel in the Setting of Type 2 Diabetes Mellitus (T2DM) and Coronary Artery Disease (CAD)
Brief Title: Impact of Chronic Kidney Disease on Clopidogrel Effects in Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Scott R. MacKenzie Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201801870 -A
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Disease (CKD); Type 2 Diabetes Mellitus (T2DM); Coronary Artery Disease (CAD)
Keywords: pharmacodynamics (PD); pharmacokinetic (PK); clopidogrel
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetes Mellitus patients with Chronic Kidney Disease (Experimental): Patients with CKD will be administered a 600-mg LD of Clopidogrel followed by a single 75-mg MD administered after 24 hours.
  Blood samples collected at baseline will be incubated with clopidogrel active metabolite.
  Interventions: Drug: Clopidogrel; Drug: Clopidogrel active metabolite
- Diabetes Mellitus patients without Chronic Kidney Disease (Active Comparator): Patients without CKD will be administered a 600-mg LD of Clopidogrel followed by a single 75-mg MD administered after 24 hours.
  Blood samples collected at baseline will be incubated with clopidogrel active metabolite.
  Interventions: Drug: Clopidogrel; Drug: Clopidogrel active metabolite

INTERVENTIONS:
Drug: Clopidogrel — Both CKD and Non-CKD patients will be administered a 600-mg LD of clopidogrel followed by a single 75-mg MD administered after 24 hours.
  Other Names: Plavix
Drug: Clopidogrel active metabolite — In both CKD and Non-CKD patients, blood samples collected at baseline only (before clopidogrel LD administration) will be incubated with escalating concentrations of clopidogrel active metabolite (1, 3 and 10 μM)
  Other Names: Plavix

SUMMARY:
Patients with diabetes mellitus (DM) and chronic kidney disease (CKD) are at increased risk of atherothrombotic events. Clopidogrel is the most widely used platelet P2Y12 receptor inhibitor in patients with coronary artery disease (CAD). However, despite its benefits, many patients still experience recurrent atherothrombotic events. The proposed study will test the central hypothesis that in DM patients the presence of CKD reduces clopidogrel-mediated P2Y12 inhibitory effects through synergistic mechanisms, which include upregulation of the P2Y12 signaling pathway and impaired clopidogrel metabolism.

DETAILED DESCRIPTION:
Patients with diabetes mellitus (DM) and coexisting chronic kidney disease (CKD) are at increased risk of atherothrombotic events, underscoring the importance of secondary prevention antiplatelet therapy in these high-risk patients. Clopidogrel is the most widely used platelet P2Y12 receptor inhibitor in patients with coronary artery disease (CAD). However, despite its clinical benefits, many patients still experience recurrent atherothrombotic events. This is in part due to the impaired effects of clopidogrel in DM patients, particularly among those with coexisting CKD. However, underlying mechanism(s) leading to magnification of impaired clopidogrel response among DM patients with CKD remain unexplored. The ever growing prevalence of CKD in patients with DM and their high risk of recurrent events underscores the need to define such mechanism(s) as this may set the basis for identifying treatment regimens leading to more effective platelet inhibition and cardiovascular protection in these high-risk patients. The proposed study will test the central hypothesis that in DM patients the presence of CKD reduces clopidogrel-mediated P2Y12 inhibitory effects through synergistic mechanisms, which include upregulation of the P2Y12 signaling pathway and impaired clopidogrel metabolism. Comprehensive pharmacokinetic and pharmacodynamic assessments, including ex vivo and in vitro experiments, evaluating the impact of CKD on antiplatelet drug response in DM patients are proposed.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM, defined according to ADA definition, on treatment with oral hypoglycemic agents and/or insulin
* Angiographically documented CAD
* On treatment with low-dose aspirin (81mg/day) for ≥30 days as part of standard of care.

Exclusion Criteria:

* Use of any antiplatelet therapy (except aspirin) in prior 30 days
* Use of parenteral or oral anticoagulation
* Active bleeding
* High risk of bleeding
* Clinical indication to be on a P2Y12 receptor inhibitor
* End-stage renal disease on hemodialysis
* Any active malignancy
* Platelet count < 100x106/µl
* Hemoglobin <9 g/dl
* Severe known liver disease
* Hemodynamic instability
* Known allergy to clopidogrel
* Pregnant / lactating females (women of childbearing age must use reliable birth control).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Franchi, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ortega-Paz L, Franchi F, Rollini F, Galli M, Been L, Ghanem G, Shalhoub A, Ossi T, Rivas A, Zhou X, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Mahowald MK, Langaee T, Jakubowski JA, Cavallari LH, Angiolillo DJ. Clopidogrel-Mediated P2Y12 Inhibition According to Renal Function in Patients With Diabetes Mellitus and CAD. JACC Basic Transl Sci. 2024 Mar 25;9(7):865-876. doi: 10.1016/j.jacbts.2024.03.003. eCollection 2024 Jul. PMID 39170956

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetes Mellitus Patients With Chronic Kidney Disease: Patients with CKD will be administered a 600-mg LD of Clopidogrel followed by a single 75-mg MD administered after 24 hours.
  Blood samples collected at baseline will be incubated with clopidogrel active metabolite.
  Clopidogrel: Both CKD and Non-CKD patients will be administered a 600-mg LD of clopidogrel followed by a single 75-mg MD administered after 24 hours.
  Clopidogrel active metabolite: In both CKD and Non-CKD patients, blood samples collected at baseline only (before clopidogrel LD administration) will be incubated with escalating concentrations of clopidogrel active metabolite (1, 3 and 10 μM)
- Diabetes Mellitus Patients Without Chronic Kidney Disease: Patients without CKD will be administered a 600-mg LD of Clopidogrel followed by a single 75-mg MD administered after 24 hours.
  Blood samples collected at baseline will be incubated with clopidogrel active metabolite.
  Clopidogrel: Both CKD and Non-CKD patients will be administered a 600-mg LD of clopidogrel followed by a single 75-mg MD administered after 24 hours.
  Clopidogrel active metabolite: In both CKD and Non-CKD patients, blood samples collected at baseline only (before clopidogrel LD administration) will be incubated with escalating concentrations of clopidogrel active metabolite (1, 3 and 10 μM)
Period: Overall Study
Arm/Group | Diabetes Mellitus Patients With Chronic Kidney Disease | Diabetes Mellitus Patients Without Chronic Kidney Disease
Started | 31 | 30
Completed | 29 | 30
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Patient with diabetes and stable coronary artery disease not on a P2Y12 inhibitor.
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Mellitus Patients With Chronic Kidney Disease | Diabetes Mellitus Patients Without Chronic Kidney Disease | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 17 | 26
  >=65 years | 22 | 13 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (10.8) | 65.2 (6.8) | 66.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 15 | 24
  White | 21 | 15 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61
Prior myocardial infarction [Count of Participants; unit: Participants] | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Index (PRI) Assessed by VASP. The Cutoff for High Platelet Reactivity is >50%
Description: Comparison of platelet reactivity measured as PRI assessed by VASP after a 600 mg clopidogrel LD between DM patients with and without CKD
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: PRI%
Arm/Group | Diabetes Mellitus Patients With Chronic Kidney Disease | Diabetes Mellitus Patients Without Chronic Kidney Disease
Number analyzed (Participants) | 29 | 30
PRI% | 67.5 (27.4) | 67.2 (30.2)

2. Secondary Outcome: Clopidogrel Active Metabolite Concentration
Description: Comparison of clopidogrel active metabolite plasma concentrations by means of AUC
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: ng*h/mL
Arm/Group | Diabetes Mellitus Patients With Chronic Kidney Disease | Diabetes Mellitus Patients Without Chronic Kidney Disease
Number analyzed (Participants) | 29 | 30
ng*h/mL | 47.1 [32.8 to 62.7] | 39.6 [19.8 to 85.8]

3. Other Pre Specified Outcome: P2Y12 Reaction Units (PRU) Assessed by VerifyNow. The Cutoff for High Platelet Reactivity is >208.
Description: Comparison of platelet reactivity measured as PRU assessed by VerifyNow after a 600 mg clopidogrel LD between DM patients with and without CKD
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Diabetes Mellitus Patients With Chronic Kidney Disease | Diabetes Mellitus Patients Without Chronic Kidney Disease
Number analyzed (Participants) | 29 | 30
PRU | 164 (91) | 156 (92)

4. Other Pre Specified Outcome: Platelet Reactivity Index (PRI) Assessed by VASP. The Cutoff for High Platelet Reactivity is >50%
Description: Comparison of of platelet reactivity measured as PRI assessed by VASP after incubation with clopidogrel active metabolite between DM patients with and without CKD
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: PRI%
Arm/Group | Diabetes Mellitus Patients With Chronic Kidney Disease | Diabetes Mellitus Patients Without Chronic Kidney Disease
Number analyzed (Participants) | 29 | 30
PRI% | 92.7 (5.6) | 94.4 (3.5)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Diabetes Mellitus Patients With Chronic Kidney Disease | Diabetes Mellitus Patients Without Chronic Kidney Disease
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT03774394/Prot_001.pdf